CLINICAL TRIAL: NCT00828542
Title: Safety of the Etonogestrel-releasing Implant During the Puerperium of Healthy Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Milena Bastos Brito, MD, PhD, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HCRP4432/2007
Record Dates: First submitted 2009-01-23; First posted 2009-01-26 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Breastfeeding; Contraception
Keywords: Adverse Effects; Etonogestrel; Postpartum period; Contraception; Hemostasis; Metabolism
MeSH Terms: conditions — Breast Feeding | interventions — etonogestrel; Medroxyprogesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- etonogestrel implant (Experimental): Etonogestrel releasing contraceptive implant (Implanon®, NV Organon, Oss, The Netherlands) inserted 24-48 h after delivery. It is compounded by 68mg of etonogestrel, 3years of duration.
  Interventions: Drug: etonogestrel implant
- depot medroxyprogesterone acetate (Active Comparator): At the 6th week postpartum, this group received intramuscular 150 mg of depot medroxyprogesterone acetate (Contracept®, EMS Sigma Pharma, Hortolandia, Brazil).
  Interventions: Drug: depot medroxyprogesterone acetate

INTERVENTIONS:
Drug: etonogestrel implant — Etonogestrel-releasing subdermal implant (Implanon) inserted during the immediate postpartum period (from 24 to 48 hours postpartum)
  Other Names: Implanon, Etonogestrel implant
  Arms: etonogestrel implant
Drug: depot medroxyprogesterone acetate — 150 mg medroxyprogesterone administered I.M. every three months starting 6 weeks after delivery
  Other Names: medroxyprogesterone
  Arms: depot medroxyprogesterone acetate

SUMMARY:
The purpose of this study to assess the safety of the etonogestrel-releasing subdermal implant (Implanon) inserted during the immediate puerperium of healthy women.

DETAILED DESCRIPTION:
Many contraceptive methods are currently available. However, about 50% of all pregnancies in the world are not planned, most of them occurring in developing countries. Long-lasting reversible contraceptives such as the etonogestrel implant represent an option for the reduction of unwanted pregnancies, especially among patients at risk for a short intergestational period. In addition to preventing an undesired pregnancy, these methods have an impact on the reduction of the maternal-fetal morbidity-mortality known to be associated with these short intervals, also minimizing the malnutrition and the cycle of poverty caused by multiparity.

On the basis of inclusion and exclusion criteria, we will selected 40 puerperae aged 18 to 35 years at the Low Risk Prenatal Care Program of the University Hospital of Ribeirão Preto, University of São Paulo (HC-FMRP). The subjects will be randomized to two types of treatment (etonogestrel-releasing implant to be inserted 24 to 48 hours after delivery or 150 mg medroxyprogesterone administered every three months starting 6 weeks after delivery). Blood samples (40 mL) will be collected in a single procedure from these patients and stored for later determination of multiple hemostatic and metabolic variables at 24-48 hours and at 6 and 12 weeks after delivery. Data on maternal and neonatal clinical parameter will be also collected.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 35 years
* Postpartum contraception desire

Exclusion Criteria:

* smoking, alcoholism or drug addiction
* presence of systemic diseases (diabetis melittus, cardiovascular disease, autoimmune diseases, liver disease, thyroid disease, or congenital renal hyperplasia)
* having a body mass index ≥ 30 kg/m2
* personal history of arterial or venous thrombosis
* using any medication that might interfere with blood coagulation or with the assessment of haemostatic and inflammatory variables
* presenting alterations in hepatic enzymes
* being allergic to local anaesthetics (xylocaine)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2007-07; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolina S Vieira, MD, PhD, Principal Investigator — University of Sao Paulo; Milena B Brito, MD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brito MB, Ferriani RA, Quintana SM, Yazlle ME, Silva de Sa MF, Vieira CS. Safety of the etonogestrel-releasing implant during the immediate postpartum period: a pilot study. Contraception. 2009 Dec;80(6):519-26. doi: 10.1016/j.contraception.2009.05.124. Epub 2009 Jul 10. PMID 19913145
- [Result] Brito MB, Ferriani RA, Meijers JC, Garcia AA, Quintana SM, Silva de Sa MF, Vieira CS. Effects of the etonogestrel-releasing contraceptive implant inserted immediately postpartum on maternal hemostasis: a randomized controlled trial. Thromb Res. 2012 Sep;130(3):355-60. doi: 10.1016/j.thromres.2012.03.029. Epub 2012 Apr 28. PMID 22542366

RESULTS

PARTICIPANT FLOW:
Groups:
- Etonogestrel Implant: Immediately after giving birth, women randomized to etonogestrel implant group had an Etonogestrel releasing contraceptive implant (Implanon®, NV Organon, Oss, The Netherlands) inserted 24-48 h after delivery. It is a long-acting reversible contraceptive method, compounded by 68mg of etonogestrel, 3years of duration.
- Depot Medroxyprogesterone Acetate: Women randomized to depot medroxyprogesterone acetate group had at the 6th week postpartum, 150 mg of depot medroxyprogesterone acetate intramuscular (Contracept®, EMS Sigma Pharma, Hortolandia, Brazil). A new injection was applied every 90 days if the patient wished to keep using the method.
Period: Overall Study
Arm/Group | Etonogestrel Implant | Depot Medroxyprogesterone Acetate
Started | 23 | 23
Completed | 20 | 20
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Etonogestrel Implant: Twenty women were allocated to receive the ETGreleasing contraceptive implant (Implanon®, NV Organon, Oss, The Netherlands) inserted 24-48 h after delivery
- Depot Medroxyprogesterone: 20 women received no contraceptives during the first 6 weeks after delivery, and at the 6th week, this group received IM 150 mg of DMPA (Contracept®, EMS Sigma Pharma, Hortolândia, Brazil)
- Total: Total of all reporting groups
Arm/Group | Etonogestrel Implant | Depot Medroxyprogesterone | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 23 | 46
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.5 (2.5) | 22.9 (4.4) | 22.6 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: Etonogestrel-releasing Contraceptive Subdermal Implant Inserted During the Immediate Puerperium Effects on the Hemostatic System of Healthy Women Over a Period of Twelve Weeks
Description: Activated protein C (APC) resistance is the most important marker of coagulation system in women using hormonal contraceptive methods.
  APC resistance was determined by testing the effect of APC on the endogenous thrombin potential (ETP) using the Calibrated Automated Thrombogram® (CAT) assay. The sensitivity ratio or APC (APCsr) of each plasma sample was determined in the presence or absence of approximately 4 nM APC (Enzyme Research Laboratories, Swansea, United Kingdom). The APC concentration was adjusted to maintain the residual thrombin generation activity in normal pooled plasma at approximately 10%. Normal pooled plasma was run in parallel on each plate.
  The normalized ratio (nAPCsr) was determined by dividing the APCsr of an individual sample by the APCsr of the pooled plasma.
  Thus, nAPCsr >1.0 indicated APC resistance.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Depot Medroxyprogesterone: 20 women received no contraceptives during the first 6 weeks after delivery, and at the 6th week, this group received IM 150 mg of depot medroxyprogesterone (Contracept®, EMS Sigma Pharma, Hortolandia, Brazil)
Arm/Group | Etonogestrel Implant | Depot Medroxyprogesterone
Number analyzed (Participants) | 20 | 20
ratio | 5.9 (1.8) | 5.5 (1.5)

2. Secondary Outcome: Maternal (Clinical and Metabolic) and Neonatal (Clinical) Safety Regarding the Use of the Etonogestrel Implant During the Immediate Postpartum Period and the First 12 Weeks Postpartum
Description: Evaluation during the immediate postpartum period was performed at the hospital 24-48 h after delivery, in the morning and after a 12-h fast. Women and newborns were both weighed (Kg), and the blood pressure (mmHg), waist circumference (WC) (cm) and height (m) of the women were each measured by the same observer. Peripheral blood samples (20 mL) were collected and processed within 2 h after being collected. After clotting the serum, samples were centrifuged at room temperature for 10 min, and the sera were stored at -80°C until they were used for the simultaneous determination of all variables except for the complete blood count, which was performed before clotting. The following variables were analyzed: fasting serum glucose; total cholesterol (TC), high density lipoprotein (HDL) cholesterol, and triglycerides (TG), and low density lipoprotein (LDL) cholesterol
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Description: No patient experienced serious adverse event as hemorrhagic or thrombotic events. The most common adverse effect reported was headache during the first three months.
Groups:
- Depot Medroxyprogesterone: 20 women received no contraceptives during the first 6 weeks after delivery, and at the 6th week, this group received IM 150 mg of depot medroxyprogesterone (Contracept®, EMS Sigma Pharma, Hortolândia, Brazil)
Arm/Group | Etonogestrel Implant | Depot Medroxyprogesterone
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 9/20 | 2/20
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etonogestrel Implant (N=20) | Depot Medroxyprogesterone (N=20)
headache (Nervous system disorders) | 9 | 2 — The most frequently reported side effect was headache [45% (9/20) vs. 10% (2/20), for the implant vs. depot medroxyprogesteone group, p=.03].

LIMITATIONS AND CAVEATS:
Patients were not blinded to treatment. However, this was not possible because the ENG group received a subdermal contraceptive implant, whereas, for ethical reasons, the control group could not receive a placebo implant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No